CLINICAL TRIAL: NCT03880214
Title: Cross Sectional Study Estimating the Prevalence and Predicting Risk Factors for Developing Chronic Oral Graft Versus Host Disease in Pediatric Patients Subjected to Hematopoietic Stem Cells Transplantation
Brief Title: Prevalence of Chronic Oral Graft Versus Host Disease Risk Factors in Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: yasmeen magdi sholkamy (Other)
Responsible Party: Sponsor-Investigator, yasmeen magdi sholkamy, principle investigator , oral medicine department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: developing chronic oral GVHD
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Oral Disease; Graft-versus-host-disease; Stem Cell Transplant Complications; Pediatric Disorder
Keywords: oral GVHD; Pediatric
MeSH Terms: conditions — Mouth Diseases; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stem cells transplanted pediatric patients: screen pediatric patients at least 3 months after they undergo allogeneic hematopoietic stem cells transplantation to detect any risk factors for developing oral manifestations of chronic graft -versus-host disease during this period

SUMMARY:
our aim is estimating the Prevalence and predicting risk factors for developing chronic oral graft versus host disease in pediatric patients subjected to hematopoietic stem cells transplantation

DETAILED DESCRIPTION:
The study will be held in Children's Cancer Hospital Egypt for pediatric patients who underwent bone marrow transplantation.

this study describes oral conditions, detect possible oral pathological manifestations and evaluate their prevalence as well as correlating it to assumed risk factor as age, sex, type of the transplant , previous acute attack of graft versus host disease and other organ involvement . A standardized Transplant Database Questionnaire will be completed Clinical examination will be performed then findings will be recorded for oral mucosal lesions , salivary flow rate in milliliter , mouth opening in milliimeter.

Sample size estimation :

The aim of this study is to screen pediatric patients at least three months after they undergo allogeneic hematopoietic stem cells transplantation to detect any risk factors for developing oral manifestations of chronic graft versus host disease during this period. Every patient fulfilling inclusion criteria in the hospital will be recruited consecutively in a period of six months starting from April 2019.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients aged between 3 and 13 who underwent bone marrow transplantation at least 3 months ago.
2. Neoplastic or non- neoplastic diseases.
3. Patient receiving any protocol of GVHD prophylactic treatment.

Exclusion Criteria:

1. Patients who do not approve to join the study.
2. Patient receiving chemo or radiotherapy .

Ages: 3 Years to 13 Years | Sex: All
Age Groups: Child
Study Population: pediatric patients at least 3 months after they undergo allogeneic hematopoietic stem cells transplantation to detect any risk factors for developing oral manifestations of chronic graft -versus-host disease during this period. Every patient fulfilling inclusion criteria in 57357 pediatric hospital will be recruited consecutively in a period of 6 months starting from.....
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
oral mucosal alterations - Comprehensive intraoral clinical examination for the soft tissue under good lightening condition to detect any abnormalities (yes/no) | 10 minutes
  Clinical examination
  - Comprehensive intraoral clinical examination for the soft tissue under good lightening condition to detect any abnormalities (yes/no) .

SECONDARY OUTCOMES:
salivary gland function | 10 minutes
  resting and stimulated saliva flow examination
sclerotic disease assessed | 2 minutes
  inter incisional distance

CONTACTS AND LOCATIONS:
Overall Officials: basma abd el alim, Study Chair — Lecturer at Department of Oral Medicine and periodontology Cairo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] (Study Result )Hull K, Oral Long-Term Complications of AllogeneicHematopoietic Stem Cell Transplantation. 2009, Doctorate degree, University of Sydney, Australia (Study Result )Müller I, van Waes H, Langerweger C, Luciano C, Rotraud K Saurenmann.Maximal mouth opening capacity: percentiles forhealthy children 4-17 years of age.Pediatric Rheumatology 2013; 11:17.